CLINICAL TRIAL: NCT03961919
Title: Evaluation of Safety and Efficacy of Treosulfan-cytarabine-fludarabine (FLAT) Combination Prior to Autologous Stem Cell Transplant (HSCT) in Elderly Patients With Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS)
Brief Title: Phase II Trial in Elderly Patients With AML or MDS in Complete Remission Not Eligible for Allogenic Transplant
Acronym: FLAT-Auto
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ciceri Fabio (Other)
Responsible Party: Sponsor-Investigator, Ciceri Fabio, Head of Hematology and Translplant Unit, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-000664-16
Record Dates: First submitted 2019-05-22; First posted 2019-05-23 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes; Transplant-Related Hematologic Malignancy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — fludarabine; Cytarabine; treosulfan; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FLAT-Auto (Experimental): Treosulfan in a combination regimen with ARA-C and fludarabine as conditioning therapy prior to autologous PBSCT
  Interventions: Drug: Fludarabine; Drug: ARA-C; Drug: Treosulfan; Procedure: Peripheral Blood Stem Cell Transplant

INTERVENTIONS:
Drug: Fludarabine — Fludarabine i.v. 30 mg/m²/d day -6 to -2
Drug: ARA-C — Cytarabine i.v. 2 g/m²/d day -6 to -2
Drug: Treosulfan — Treosulfan i.v. 10 g/m²/d day -6 to -4
Procedure: Peripheral Blood Stem Cell Transplant — Autologous stem-cell transplantation i.v.: day 0 (source: peripheral blood)
  Pegylated-Filgrastim s.c. 6 mg day +3

SUMMARY:
FLAT-Auto is a phase II trial. fludarabine and ARA-C will be combined with the alkylating agent treosulfan (FLAT), to investigate the feasibility and the efficacy of a new regimen, supported with autologous peripheral blood SCT (PBSCT), as final postremission consolidation in AML/MDS elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Pts with de novo or secondary AML or with Int 2 or High risk MDS according to IPSS.
* Pts unable or unfit to receive SCT from an HLA (human leukocyte antigen)-identical related (SIB) or unrelated (MUD), or HLA-haploidentical related (HAPLO) donor.
* Hematologic CR (Appendix D) after 1 or 2 cycles of induction standard chemotherapy.
* Successful collection of autologous PBSC: ≥ 5.0x10e6 /kg patient bodyweight (BW)
* Age ≥ 65 years.
* Performance status 0-2 ECOG (Eastern Cooperative Oncology Group), 60-100% Karnofsky (Appendix E).
* Written informed consent.

Exclusion Criteria:

* Diagnosis of AML M3.
* Second concomitant malignancies.
* Severe concomitant illnesses/medical conditions (e.g. impaired respiratory and/or cardiac function).
* Known and manifested malignant involvement of the central nervous system (CNS)
* Active infectious disease
* HIV- positivity or active hepatitis infection
* Impaired liver function (bilirubin > 1.5 x upper normal limit; transaminases > 3.0 x upper normal limit)
* Impaired renal function (creatinine-clearance < 60 ml/min; serum creatinine > 1.5 x upper normal limit).
* Known hypersensitivity to treosulfan and/or cytarabine and/or fludarabine
* Participation in another experimental drug trial within 4 weeks before day -6
* Non-cooperative behaviour or non-compliance
* Psychiatric diseases or conditions that might impair the ability to give informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-02-10 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of disease free survival from first Complete Remission (CR) | 2 years after transplantation
  Evaluation of disease-free survival (DFS) duration from documented first CR of AML or MDS with intermediate 2 or high IPSS (International Prognostic Score System).

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Ciceri, MD, Principal Investigator — San Raffaele Hospital IRCCS
Locations (1):
- Ospedale San Raffaele, Milan, Lombardy, Italy